CLINICAL TRIAL: NCT05712369
Title: Phenotype and Function of Reconstituting B-cells in Steroid Dependent or Frequently Relapsing Nephrotic Syndrome After B-cell Depletion: Insight Into the Disease Pathogenesis and Identification of Predictors of Relapse
Brief Title: B Cells in Idiopathic Nephrotic Syndrome
Acronym: BLADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLADE
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic syndrome; Steroids, B cells; B cells; Anti-CD20 antibodies
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prospective cohort (Experimental): Patients with INS due to biopsy-proven MCD or FSGS or MesGN candidate to anti-CD20 monoclonal antibodies therapy.
  Interventions: Other: Blood sampling
- Retrospective cohort (Experimental): Patients with INS due to biopsy-proven MCD or FSGS or MesGN, treated with anti-CD20 monoclonal antibodies therapy.
  Interventions: Other: Blood sampling
- Healthy volunteers cohort (Active Comparator): Subjects not known to suffer of any significant illness, not assuming any medication or drug on a regular basis.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Before the anti-CD20 monoclonal antibodies treatment (e.g. Rituximab/Ofatumumab) and after 6, 9 and 12, 24 months from the first infusion the following blood samples will be collected for the analysis of lymphocyte subpopulations:
  * 50/100 mL of blood (20 mL for pediatric patients) for Peripheral Blood Mononuclear Cells (PBMCs) isolation.
  * 8 mL of blood (both adult and pediatric) to obtain serum. Serum will be obtained by standard centrifugation and PBMC will be isolated by Ficoll-Paque® density gradient centrifugation, according to manufacturer's instruction.

SUMMARY:
The main aim of the present study is to determine whether reconstitution of different B-cell subpopulations can predict relapse after treatment with B-cell depleting antibodies in adult with NS, and whether specific B- or T-cell anomalies (as well as dysregulation of other circulating immune cell subsets) may play a role in the disease pathogenesis of SDNS and FRNS.

DETAILED DESCRIPTION:
The role of the immune system in Idiopathic Nephrotic Syndrome (INS) of Minimal Change Disease (MCD), Mesangial proliferative Glomerulonephritis (MesGN) or Focal and Segmental Glomerulosclerosis (FSGS) has been widely investigated. However, among immune cell populations, a major player in disease pathogenesis was never found.

The efficacy of B cell depleting therapy with anti-CD20 monoclonal antibodies suggests that B lymphocytes may play a pivotal role.

Preliminary data suggest that memory B cells may be the responsible of the Nephrotic Syndrome (NS) relapse after rituximab treatment in children with Steroid Dependent Nephrotic Syndrome (SDNS) or Frequently-Relapsin gnephrotic Syndrome (FRNS), enforcing the role of the B cell lineage in the disease pathogenesis.

NS is a severe glomerular disease affecting more frequently children and young adult. It is characterized by edema, heavy proteinuria and hypoalbuminemia, the clinical counterpart of the alteration of the selective glomerular permeability barrier. Despite extensive investigation, the mechanism and the immune cell population responsible for the disruption of glomerular filtration barrier and, consequently, of the development of proteinuria is still not clearly defined. However, the efficacy of the different immunosuppressive approaches including prednisone and anti-CD20 antibodies in the treatment of NS strongly suggests a central role of the immune system, in particular the role of B cells in the pathogenesis SDNS. Recent evidence indicates that, after B cell depletion, the delayed reconstitution of the switched memory B cells in children with SDNS was significantly and independently protective against relapse. These results suggest that recovery of switched memory B-cells after anti-CD20 therapies could be a useful predictor of subsequent relapse of the NS in SDNS and FRNS patients, and that memory B-cells may play a role in the pathogenesis of SDNS or FRNS in children.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children (≥6 and <18 years old) and adults.
2. Patients with biopsy-proven MCD or FSGS or MesGN candidate to (prospective cohort) or treated with (retrospective cohort) anti-CD20 monoclonal antibodies (when possible) due to INS and fulfilling the following conditions:

   * SDNS: defined as two consecutive relapses of the NS during corticosteroid therapy, or within 14 days of ceasing therapy;
   * FRNS: defined as two or more relapses within 6 months of initial response, or four or more relapses in any 12-month period; Note: relapse in pediatric patients is defined as a urinary protein to creatinine ratio > 2000 mg/g or a positive urine dipstick (≥ 3+) for 3 consecutive days; in adult is defined as a urinary protein to creatinine ratio > 3500 mg/g or by proteinuria >3.5 g/day after remission has been obtained.

   Patients will be included irrespective of previous (retrospective cohort) or planned (prospective cohort) treatments with anti-CD20 monoclonal antibodies.
   * SRNS not associated with known genetic abnormalities of the glomerular barrier consisting in persistent nephrotic-range proteinuria (no complete/partial remission) despite prednisone 1 mg/kg/day or 2 mg/kg every other day for >4 months (adults) or despite prednisone 60 mg/m2/day or 2 mg/kg/day to a maximum 60 mg/day (pediatrics), having no pathogenic mutations at the sequencing analysis for the known genes associated with NS (see appendix Table 1 for the full list of genes); Note: patients with biopsy-proven MCD/MesGN/FSGS recurrence in the kidney graft after renal transplantation with clinical features NS will be also considered.
   * SRNS due to mutations in podocyte genes consisting in persistent nephrotic-range proteinuria (no complete/partial remission) despite prednisone 1 mg/kg/day or 2 mg/kg every other day for > 4 months (adults) or despite prednisone 60 mg/m2/day or 2 mg/kg/day to a maximum 60 mg/day (pediatrics), harbouring pathogenic mutations at the sequencing analysis for genes associated with NS (see appendix Table 1for the full list of genes). This last condition will not consider possible treatments for the enrolment, as the patients usually are not treated with anti-CD20 monoclonal antibodies.
3. For adults: written informed consent according to the guidelines of the Declaration of Helsinki.
4. For children: written informed consent (according to the guidelines of the Declaration of Helsinki) of parent(s) or guardian.

Healthy volunteers Healthy subjects (>18 years) not known to suffer of any significant illness, not assuming any medication or drug on a regular basis, and whose mental state is such that they are able to understand and give valid consent to the study will be recruited among researchers and personnel of the IRCSS - Mario Negri Institute for Pharmacological Research. Only healthy subjects with negative urine analysis (urine dipstick, multistick will be considered for this study.

Exclusion Criteria:

1. Reasonable possibility of a secondary cause of NS: active hepatitis B or C infection, or other chronic systemic infections; malignancy; drug abuse.
2. Legal incapacity, intellectual disability/mental retardation, dementia, uncooperative attitude or any other evidence that patient will not be able to understand the study procedures and aims and to give written informed consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in frequency of circulating B cell subpopulations | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in frequency of circulating T cell | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in NK-cell | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in monocyte | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in dendritic cell subpopulations | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in serum levels of cytokines | At baseline, 6,9 12 and 24 months after treatment.
Differences between NS patients who relapse (R) or who achieved sustained remission (NR) after B-cell depleting monoclonal antibody treatment in serum levels of immunoglobulin classes and subclasses | At baseline, 6,9 12 and 24 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No